CLINICAL TRIAL: NCT00006270
Title: Study of the Approximate Entropy of Adrenocorticotropic Hormone and Cortisol Secretion in Patients With Head Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Other Study IDs: 199/15376; UTMB-98-018; UTMB-GCRC-486
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Brain Injury; Craniocerebral Trauma
Keywords: brain injury; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Cosyntropin; Metyrapone

INTERVENTIONS:
Drug: cosyntropin
Drug: metyrapone

SUMMARY:
OBJECTIVES: I. Determine the randomness of adrenocorticotropic hormone (ACTH) and cortisol secretion using approximate entropy in patients who have sustained a head injury.

II. Determine the correlation between randomness of ACTH and cortisol secretion and stages of sleep in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are stratified according to type of injury (closed head injury due to trauma vs vascular accidents). Patients are admitted two times for overnight assessment.

Admission 1: Patients receive cosyntropin IV. Blood is drawn at 30 and 60 minutes after IV infusion. Patients receive oral metyrapone before sleep. A sham sleep study is conducted through the night and patients' blood is drawn in the morning.

Admission 2: At least 2 weeks after admission 1, patients return for an overnight admission. Starting in the evening, blood is drawn every 15 minutes for 12 hours. A sleep study is conducted through the night.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Patients who have sustained head injury

Closed head injury from trauma OR

Vascular accidents like strokes and hemorrhages

--Prior/Concurrent Therapy--

Endocrine therapy: No concurrent cortisol replacement

Other: No blood donation during and for 1 month after study

--Patient Characteristics--

Hematopoietic: Hemoglobin normal

Other:

* No hypopituitarism
* No body mass index of 28 or greater
* Not pregnant or nursing
* Must have normal menstrual cycles
* No severe mental impairment
* Must not require legal guardian

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32
Dates: Start 1998-02

CONTACTS AND LOCATIONS:
Overall Officials: Randall Urban, Study Chair — University of Texas
Locations (2):
- United States (2):
  - Transitional Learning Community, Galveston, Texas
  - University of Texas Medical Branch, Galveston, Texas